CLINICAL TRIAL: NCT00211614
Title: Proton Pump Inhibitor Therapy for Mild to Moderate Obstructive Sleep Apnea
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No enrollment.
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Dennis Auckley, MD, MD, MetroHealth Medical Center
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: IRB04-00029
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Obstructive Sleep Apnea; Gastroesophageal Reflux
Keywords: Obstructive Sleep Apnea; Gastroesophageal Reflux; Proton Pump Inhibitor; Lansoprazole (Prevacid); Quality of Life
MeSH Terms: conditions — Sleep Apnea, Obstructive; Gastroesophageal Reflux | interventions — Lansoprazole

INTERVENTIONS:
Drug: Lansoprazole

SUMMARY:
Obstructive Sleep Apnea (OSA) is common in modern society, affecting up to 5% of working middle-aged adults in the United States. Obesity is the number one risk factor for the development of OSA. Consequences of untreated OSA are varied and significant and included numerous neuropsychiatric parameters such as mood alterations, depression, anxiety, diminished social interactions, and decreased quality of life. Mounting evidence suggests that treatment of OSA can improve many of these outcomes. The primary treatment modality for this condition is continuous positive airway pressure (CPAP). This device delivers positive pressure to the upper airway in order to prevent its collapse during sleep. Unfortunately, many patients do not choose to use CPAP or have difficulty with these devices. This results in many individuals with OSA either going without therapy or unable to reap the full benefits of treatment.

Gastroesophageal reflux (GERD) is also common in the United States and may, in some instances, be directly related to weight gain. Survey studies have suggested that symptomatic GERD is more common in patients with OSA. Whether there exists a cause and effect relationship between these two conditions is not known at present. It has been suggested that GERD may contribute to OSA by narrowing the upper airway.

This study will examine the effect of treatment of GERD on mild to moderate OSA. Fifty individuals identified as having mild to moderate OSA (diagnosed by overnight sleep study or PSG) and GERD (confirmed by an esophageal probe) will be enrolled. Both men and women will be included in this study and no "special populations" will be utilized. Subjects will fill out questionnaires to subjectively measure sleepiness, OSA-related symptoms, GERD-related symptoms, and sleep apnea-related quality of life. They will then be randomized to receive either 12 weeks of the proton pump inhibitor lansoprazole (Prevacid) or placebo (twenty five subjects per group). Upon completion of the 12 week trial, subjects will return and the following data will be collected; repeat all of the baseline questionnaires, repeat PSG and repeat pH probe.

Results from this study will help to establish the relative effectiveness of a novel form of therapy for a common yet difficult to manage medical condition. . The risks to subjects enrolled in the study are minimal and therefore the benefit to risk ratio is heavily in favor of performing the study.

DETAILED DESCRIPTION:
See above.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (> 18 years old) with mild to moderate OSA (as defined by an apnea-hypopnea index between 5 and 30) currently on no therapy.
2. GERD as documented by 24 pH probe (> 6% of the time with pH < 4).
3. Agreeable to participating in the study

Exclusion Criteria:

1. Those not meeting the inclusion criteria
2. Prisoners, minors, incompetent subjects, unconscious subjects, house staff and students, pregnant women
3. Oxygen dependent, requiring supplemental oxygen during sleep, or significant hypoxia during the initial PSG (O2 sats < 85% for > 5 minutes of sleep)
4. Severe cardiac or pulmonary disease (CHF with EF < 40%, active coronary ischemia or unstable angina, uncontrolled arrythmias,COPD or other lung condition requiring supplemental oxygen or documented hypercapnia of a pCO2 > 45).
5. Neuromuscular disease with hypercapnia (pCO2 > 45)
6. Any cancer with a prognosis of < 1 year survival
7. Use of H2 blocker therapy or PPI therapy within 14 days of the initial PSG.
8. Individuals requiring routine use of sleep aids (i.e. benzodiazepines or other sedatives)
9. Individuals with active alcohol or substance abuse
10. Night shift workers or those working rotating shifts
11. Disabling sleepiness (Epworth Sleepiness Scale > 17 or history of accidents related to sleepiness) that places individual at risk for accidents.
12. Inability to complete study questionnaires
13. Allergy to lansoprazole

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-07 (Estimated); Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Reduction in the apnea-hypopnea index

SECONDARY OUTCOMES:
Numerous sleep parameters (arousals, sleep efficiency, sleep architecture), daytime sleepiness, GERD sxs, QOL measures

CONTACTS AND LOCATIONS:
Overall Officials: Dennis H Auckley, MD, Principal Investigator — MetroHealth Medical Center (Case Western Reserve University)
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States